CLINICAL TRIAL: NCT03957616
Title: Incidence of Paraneoplastic Neurological Syndromes and Autoimmune Encephalitis in France Between 2016 and 2018
Brief Title: Incidence of Paraneoplastic Neurological Syndromes and Autoimmune Encephalitis
Acronym: IPNSAE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: IPNSAE
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Paraneoplastic Neurological Syndrome; Autoimmune Encephalitis
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Paraneoplastic neurological syndromes patients: Patients tested for Paraneoplastic neurological syndromes (PNS) and Autoimmune Encephalitis (AE) with a lumbar puncture, with detection of an antibody or negative, but with PNS clinically diagnosed.

SUMMARY:
This study aims to provide an estimate of the incidence of paraneoplastic neurological syndromes and autoimmune encephalitides in France between the years 2016 and 2018. The study will describe the incidence of antibody subtypes and regional variations.

ELIGIBILITY:
Inclusion Criteria:

- Clinical diagnosis of Paraneoplastic Neurological Syndrome (PNS) or Autoimmune Encephalitis (AE) made by the referring physician to the national center for PNS and AE in Lyon between 2016 and 2018

Exclusion Criteria:

* Data on location of diagnosis missing
* Patients diagnosed out of the mainland French territory
* Patients for whom insufficient data was available

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with a paraneoplastic neurological syndrome or autoimmune encephalitis in France and referred to the national center in Lyon between 2016 and 2018.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-05-30 (Estimated); Primary Completion 2019-05-30 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and prevalence of diagnosed Paraneoplastic Neurological Syndromes (PNS) and Autoimmune Encephalitis (AE) between 2016 and 2018. | 3 years
  Comparison between general population of the French counties and the cohort of PNS to calculate incidence and prevalence.

SECONDARY OUTCOMES:
Location (city) of diagnosis | 1 hour
  Name of city where the diagnosis of Paraneoplastic Neurological Syndromes (PNS) or Autoimmune Encephalitis (AE) was made.
French general population of each counties | 3 years
  Person years for each region

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme Honnorat, Principal Investigator — center for paraneoplastic neurological syndromes and autoimmune encephalitis
Locations (1):
- Centre de référence des syndromes neurologiques paranéoplasiques et encéphalites auto-immunes, Lyon, France